CLINICAL TRIAL: NCT00776477
Title: The Clopidogrel and Aspirin After Surgery for Coronary Artery Disease
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: China National Center for Cardiovascular Diseases (Other Government)
Responsible Party: shengshou hu,MD, Institute of cardiovascular diseases& Fuwai Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCCD20080101
Record Dates: First submitted 2008-10-19; First posted 2008-10-21 (Estimated); Last update posted 2008-10-21 (Estimated); Status verified 2008-10

CONDITIONS: Atherosclerosis
MeSH Terms: conditions — Atherosclerosis | interventions — Clopidogrel; Aspirin

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: clopidogrel and aspirin
- 2 (Active Comparator)
  Interventions: Drug: aspirin

INTERVENTIONS:
Drug: clopidogrel and aspirin — clopidogrel 75mg daily and aspirin 100mg daily
  Arms: 1
Drug: aspirin — aspirin 100mg daily
  Arms: 2

SUMMARY:
Clopidogrel is a antiplatelet agent and is effective at reducing intimal hyperplasia in animal models of thrombosis.Several large clinical trials have demonstrated that clopidogrel with aspirin can reduce ischemic events and mortality in patients with atherosclerotic disease,therefore the combination of two antiplatelets might be useful to prevent patients received coronary artery bypass graft surgery from Saphenous vein graft disease. the aim of this study is to estimate the safety and efficacy of clopidogrel and aspirin therapy versus aspirin alone in patients after CABG.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing primary multi-vessel CABG with at least two saphenous vein grafts, with or without the use of cardiopulmonary bypass.

Exclusion Criteria:

* Emergency surgery
* Valve surgery
* Redo CABG
* Left ventricle ejection fraction < 30%
* Preoperative use of clopidogrel (with the exception of the current admission)
* Preoperative use of warfarin
* Allergy to aspirin or clopidogrel
* History of cerebrovascular accident
* History of severe liver disease
* Morbid obesity
* Current malignancy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2007-12; Primary Completion 2008-12 (Estimated)

PRIMARY OUTCOMES:
Vein graft patency examined by CT scan | three months after surgery

SECONDARY OUTCOMES:
Incidence of major adverse coronary events Incidence of major bleeding events | two years following surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of cardiovascular diseases,Fuwai hospital, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Gao G, Zheng Z, Pi Y, Lu B, Lu J, Hu S. Aspirin plus clopidogrel therapy increases early venous graft patency after coronary artery bypass surgery a single-center, randomized, controlled trial. J Am Coll Cardiol. 2010 Nov 9;56(20):1639-43. doi: 10.1016/j.jacc.2010.03.104. PMID 21050973